CLINICAL TRIAL: NCT02340975
Title: A Phase 1b/2 Study of MEDI4736 in Combination With Tremelimumab, MEDI4736 Monotherapy, and Tremelimumab Monotherapy in Subjects With Metastatic or Recurrent Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Phase 1b/2 Study of MEDI4736 With Tremelimumab, MEDI4736 or Tremelimumab Monotherapy in Gastric or GEJ Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00021
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Immunotherapy; Antibodies, Monoclonal; Tremelimumab; MEDI4736
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W) (Experimental): Participants in second-line therapy with gastric or gastroesophageal junction (GEJ) adenocarcinoma will receive intravenous (IV) infusion of 20 mg/kg MEDI4736 every 4 weeks (Q4W) for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, participants will receive MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
  Interventions: Biological: MEDI4736 + tremelimumab
- Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (Experimental): Participants in second-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma will receive IV infusion of 20 mg/kg MEDI4736 Q4W for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, participants will receive MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
  Interventions: Biological: MEDI4736 + tremelimumab
- Phase 2 Arm B-M10 mg/kg (Q2W) (Experimental): Participants in second-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma will receive IV infusion of 10 mg/kg MEDI4736 Q2W for 12 months (up to 26 doses).
  Interventions: Biological: MEDI4736
- Phase 2 Arm C-T10 mg/kg (Q4W) (Experimental): Participants in second-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma will receive IV infusion of 10 mg/kg tremelimumab Q4W for 7 doses and then Q12W for 2 doses for 12 months (for a total of up to 9 doses).
  Interventions: Biological: Tremelimumab
- Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (Experimental): Participants in third-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma will receive IV infusion of 20 mg/kg MEDI4736 Q4W for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, participants will receive MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
  Interventions: Biological: MEDI4736+tremelimumab
- Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (Experimental): Participants in second and third-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma and a positive IFN-γ gene expression signature will receive IV infusion of 20 mg/kg MEDI4736 Q4W for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, participants will receive MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
  Interventions: Biological: MEDI4736 + tremelimumab

INTERVENTIONS:
Biological: MEDI4736 + tremelimumab — MEDI4736 will be administered by IV infusion in combination with tremelimumab.
  Arms: Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Biological: MEDI4736 + tremelimumab — MEDI4736 will be administered by IV infusion in combination with tremelimumab.
  Arms: Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Biological: MEDI4736 — MEDI4736 will be administered by IV infusion.
  Arms: Phase 2 Arm B-M10 mg/kg (Q2W)
Biological: Tremelimumab — Tremelimumab will be administered by IV infusion.
  Arms: Phase 2 Arm C-T10 mg/kg (Q4W)
Biological: MEDI4736+tremelimumab — MEDI4736 will be administered by IV infusion in combination with tremelimumab.
  Arms: Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Biological: MEDI4736 + tremelimumab — MEDI4736 will be administered by IV infusion in combination with tremelimumab.
  Arms: Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)

SUMMARY:
This is a randomized, multicenter, open-label, dose-exploration and dose-expansion study to evaluate the safety, tolerability, antitumor activity, PK, pharmacodynamics, and immunogenicity of MEDI4736 in combination with tremelimumab, MEDI4736 monotherapy or tremelimumab monotherapy in participants with metastatic or recurrent gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants
2. 18 years and older
3. Histological or cytological confirmation of metastatic or recurrent gastric or gastroesophageal junction adenocarcinoma
4. Participants must have received and have progressed, or are refractory to standard regimens
5. Participants must have at least one lesion amenable to biospy

Exclusion Criteria:

1. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment
2. Previous immunotherapy
3. Concurrent or prior use of immunosuppressive medication with 14 days
4. Active or prior documented autoimmune or inflammatory disease within 3 years with some exceptions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, LLC MedImmune, LLC, Study Director — MedImmune LLC
Locations (22):
- United States (13):
  - Research Site, Los Angeles, California
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Research Site, Montreal, Quebec, Canada
- Japan (3):
  - Research Site, Kawasaki-shi
  - Research Site, Kōtoku
  - Research Site, Osaka
- Research Site, Singapore, Singapore
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan District

REFERENCES:
- See also: Redacted D4190C00021 SAP v3.0 final — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4190C00021&attachmentIdentifier=55b427f9-1d33-4bb5-871e-556d7cad26eb&fileName=Redacted_D4190C00021_SAP_v3.0_final.pdf&versionIdentifier=
- See also: Protocol D4190C00021_Redacted_Final_April2020_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4190C00021&attachmentIdentifier=97082c09-4d33-45f5-a36f-d61451f3915e&fileName=Protocol_D4190C00021_Redacted_Final_April2020_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States of America, Japan, Korea, Taiwan and Singapore between 31Mar2015 and 29Apr2019.
Pre-assignment Details: A total of 114 participants were randomized in the study, out of which 113 participants received study treatment.
Groups:
- Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W): Participants in second-line therapy with gastric or gastroesophageal junction (GEJ) adenocarcinoma received intravenous (IV) infusion of 20 mg/kg MEDI4736 every 4 weeks (Q4W) for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
- Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W): Participants in second-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma received IV infusion of 20 mg/kg MEDI4736 Q4W for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
- Phase 2 Arm B-M10 mg/kg (Q2W): Participants in second-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma received IV infusion of 10 mg/kg MEDI4736 Q2W for 12 months (up to 26 doses).
- Phase 2 Arm C-T10 mg/kg (Q4W): Participants in second-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma received IV infusion of 10 mg/kg tremelimumab Q4W for 7 doses and then Q12W for 2 doses for 12 months (for a total of up to 9 doses).
- Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W): Participants in third-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma received IV infusion of 20 mg/kg MEDI4736 Q4W for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
- Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W): Participants in second and third-line therapy with metastatic or recurrent gastric or GEJ adenocarcinoma and a positive IFN-γ gene expression signature received IV infusion of 20 mg/kg MEDI4736 Q4W for 4 months (up to 4 doses) in combination with IV 1 mg/kg tremelimumab Q4W for 4 months (up to 4 doses in total). Thereafter, MEDI4736 monotherapy (10 mg/kg) every 2 weeks (Q2W) to complete a total of 12 months of therapy (up to 18 additional doses).
Period: Overall Study
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W) | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Started | 6 | 27 | 24 | 12 | 25 | 19
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 27 | 24 | 12 | 25 | 19
Not completed — Death | 6 | 23 | 21 | 7 | 21 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3 | 2 | 0
Not completed — Other | 0 | 4 | 0 | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W) | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Total
Number analyzed (Participants) | 6 | 27 | 24 | 12 | 25 | 19 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.0 (12.7) | 60.4 (13.5) | 59.8 (12.0) | 52.3 (16.0) | 58.6 (10.7) | 59.9 (12.8) | 59.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 5 | 4 | 9 | 5 | 30
  Male | 6 | 20 | 19 | 8 | 16 | 14 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 27 | 23 | 12 | 25 | 18 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 7 | 11 | 5 | 12 | 13 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 20 | 13 | 6 | 13 | 6 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) in Phase 1b
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Participants
  TEAEs | 6
  TESAEs | 2

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Phase 1b
Description: A DLT was defined as any Grade 3 or higher toxicity that occurs during the DLT evaluation period (From first dose of Study drug [Day 1] through 28 days after the administration of MEDI4736 and tremelimumab). The DLTs are: any Grade 4 immune-related adverse event (irAE), any Grade >=3 non-irAE, >= Grade 3 colitis, Grade 3 or 4 noninfectious pneumonitis irrespective of duration, Grade 2 pneumonitis, liver transaminase elevation > 8 × upper limit of normal (ULN) or total bilirubin > 5 × ULN. Immune-related AEs are defined as AEs of an immune nature (ie, inflammatory) in the absence of a clear alternative etiology.
Time Frame: From first dose of Study drug (Day 1) through 28 days after the administration of MEDI4736 and tremelimumab
Population: Dose limiting toxicity (DLT) evaluable population included all participants in the Phase 1b who received the Study drug and completed safety follow-up through the DLT evaluation period or experience a DLT during the DLT evaluation period (From first dose of Study drug [Day 1] through 28 days after the administration of MEDI4736 and tremelimumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Participants | 1

3. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs in Phase 1b
Description: Number of participants with clinical laboratory abnormalities reported as TEAEs are reported. Clinical laboratory abnormalities are defined as any abnormal findings in analysis of serum chemistry, hematology, and urine.
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Participants
  Anaemia | 1
  Lymphopenia | 1
  Haemoglobin decreased | 1
  Prothrombin time prolonged | 1
  Activated partial thromboplastin time prolonged | 1
  Blood alkaline phosphatase increased | 1
  Blood bilirubin increased | 1
  Gamma-glutamyltransferase increased | 2
  Transaminases increased | 1

4. Primary Outcome: Number of Participants With Abnormal Vital Signs and Physical Examinations Reported as TEAEs in Phase 1b
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal findings in the vital signs parameters (temperature, blood pressure [BP], pulse rate [or pulse oximetry at screening], and respiratory rate). Abnormal physical examinations are defined as any abnormal impact on measurements of height and weight.
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Participants
  Pyrexia | 1
  Weight decreased | 1

5. Primary Outcome: Number of Participants With Abnormal Electrocardiograms Reported as TEAEs in Phase 1b
Description: Number of participants with abnormal electrocardiograms (ECGs) reported as TEAEs are reported. Abnormal ECGs are defined as any abnormal findings in heart rate, PR, RR, QRS and QT intervals from the primary lead of the digital 12-lead ECG.
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Participants | 1

6. Primary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline in Phase 1b
Description: The ECOG scale of performance status describes the level of functioning of participants in terms of their ability to care for themselves, daily activity, and physical ability. ECOG Performance Status Scorings are: 0= fully active, able to carry on all pre-disease performance without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (for example, light house work, office work); 2= ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3= capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5= dead. The baseline performance status of participants is presented.
Time Frame: Baseline (Day 1)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Participants
  ECOG 0 | 4
  ECOG 1 | 2

7. Primary Outcome: Percentage of Participants With Objective Response (OR) in Phase 2
Description: OR: best overall response (BOR) of confirmed complete response (CR) or partial response (PR) per RECIST v1.1. BOR: best response (CR, PR, stable disease [SD], progressive disease [PD], and not evaluable) among all overall responses recorded from date of randomization for Arm A, B, C participants or date of first dose of study drug for Arms D, E participants until progression, or last evaluable disease assessment or discontinuation from the study, whichever occurred first. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD on study; PD: at least 20% increase in SOD of target lesions from smallest sum on study (at least 5mm), appearance of one or more new lesions, substantial worsening in non-target disease, increase in tumor burden leading to discontinuation of therapy.
Time Frame: From Day 1 up to End of the Treatment (EOT), 90 days post-EOT, every 3 months (Q3M) after Day 90 post-EOT up to 12 months post-EOT, and every 6 months after month 12 post-EOT (approximately up to 4 years and one month)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Percentage of participants | 11.1 [2.4 to 29.2] | 0 [0.0 to 14.2] | 8.3 [0.2 to 38.5] | 4.0 [0.1 to 20.4] | 15.8 [3.4 to 39.6]
Statistical Analysis 1: Comparison: Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) vs Phase 2 Arm B-M10 mg/kg (Q2W); Test type: Other — Comparison; p = 0.2376, Fisher Exact; Mean Difference (Net) = 11.1, 95% CI 2-sided [-0.7 to 23.0]
Statistical Analysis 2: Comparison: Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) vs Phase 2 Arm C-T10 mg/kg (Q4W); Test type: Other — Comparison; p = 1.0000, Fisher Exact; Median Difference (Net) = 2.8, 95% CI 2-sided [-16.8 to 22.4]

8. Primary Outcome: Progression Free Survival at 6 (PFS-6) Month in Phase 2
Description: The PFS-6 is the 6-month progression-free survival rate, which was the percentage of participants who were progression free and alive at 6 months. PFS was defined as the time from the date of first dose of study drug for Arm A, B, and C participants or the date of first dose of study drug for Arm D and Arm E participants to the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1) or death due to any cause. PFS was censored at the date of their last evaluable tumor assessment. Kaplan Meier method was used to evaluate PFS-6.
Time Frame: From Day 1 upto 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Percentage of participants | 12.1 [3.1 to 27.9] | NA [NA to NA] — No participants were progression free at 6 months. | 23.3 [3.6 to 52.9] | 12.5 [3.1 to 28.7] | 5.3 [0.4 to 21.4]

9. Secondary Outcome: Percentage of Participants With Objective Response in Phase 1b
Description: OR: best overall response (BOR) of confirmed complete response (CR) or partial response (PR) per RECIST v1.1. BOR: best response (CR, PR, stable disease [SD], progressive disease [PD], and not evaluable) among all overall responses recorded from date of randomization of participants or date of first dose of study drug until progression, or last evaluable disease assessment or discontinuation from the study, whichever occurred first. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD on study; PD: at least 20% increase in SOD of target lesions from smallest sum on study (at least 5mm), appearance of one or more new lesions, substantial worsening in non-target disease, increase in tumor burden leading to discontinuation of therapy.
Time Frame: as for outcome 7
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Percentage of participants | 0 [0.0 to 45.9]

10. Secondary Outcome: Duration of Stable Disease (DSD) in Phase 1b
Description: The DSD was defined as the time from the date of first dose of study treatment for Phase 1b until the first date of documented PD (per RECIST v1.1), or death due to any cause, whichever occurred first. PD is at least a 20% increase in sum of diameters of target lesions from smallest sum on study (at least 5mm), appearance of one or more new lesions, substantial worsening in non-target disease, increase in tumor burden leading to discontinuation of therapy. Kaplan Meier method was used to evaluate DSD.
Time Frame: as for outcome 7
Population: As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received. DSD was analyzed for participants with SD.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 2
Months | 5.4 [3.5 to 7.4]

11. Secondary Outcome: Median Best Percentage Change From Baseline of the Sum of Longest Diameters (SLD) of Target Lesions in Phase 1b
Description: Best percentage change from baseline of the SLD of target lesions per RECIST v1.1 was derived as the biggest decease or the smallest increase from baseline on the SLD among all post-baseline disease assessment including unscheduled assessments. Best percent change is the maximum reduction from baseline or the minimum increase from baseline in the absence of a reduction.
Time Frame: as for outcome 7
Population: as for baseline characteristics
Measure: Median (Full Range); unit: mm
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
mm | 17.7 [-3.2 to 115.1]

12. Secondary Outcome: Percentage of Participants With Disease Control at 16 Weeks in Phase 1b
Description: The disease control rate at 16 weeks was defined as the percentage of participants who achieved a BOR of confirmed CR, confirmed PR, or had SD with duration of SD for a minimum duration of 110 days, following the date of first dose of study drug. The DC was defined as a BOR of confirmed CR, confirmed PR or SD per RECIST v1.1. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD on study.
Time Frame: From Day 1 up to 16 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Percentage of participants | 33.3 [4.3 to 77.7]

13. Secondary Outcome: Percentage of Participants With Disease Control at 24 Weeks in Phase 1b
Description: The disease control rate at 24 weeks was defined as the percentage of participants who achieved a BOR of confirmed CR, confirmed PR, or had SD with duration of SD for a minimum duration of 166 days, following the date of first dose of study drug. The DC was defined as a BOR of confirmed CR, confirmed PR or SD per RECIST v1.1. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD on study.
Time Frame: From Day 1 up to 24 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Percentage of participants | 16.7 [0.4 to 64.1]

14. Secondary Outcome: Progression Free Survival at 6 Month in Phase 1b
Description: The PFS-6 is the 6-month progression-free survival rate, which was the percentage of participants who were progression free and alive at 6 months. PFS was defined as the time from the date of first dose of study drug for Phase 1b participants to the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1) or death due to any cause. PFS was censored at the date of their last evaluable tumor assessment. Kaplan Meier method was used to evaluate PFS.
Time Frame: From Day 1 upto 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 6
Percentage of participants | 16.7 [0.8 to 51.7]

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) in Phase 2
Description: as for outcome 1
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Participants
  TEAEs | 27 | 23 | 12 | 22 | 18
  TESAEs | 14 | 16 | 10 | 15 | 12

16. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs in Phase 2
Description: as for outcome 3
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Participants
  Anaemia | 9 | 3 | 3 | 7 | 4
  Lymphocyte count decreased | 1 | 1 | 1 | 0 | 0
  White blood cell count decreased | 0 | 0 | 1 | 0 | 0
  International normalised ratio increased | 3 | 0 | 1 | 1 | 0
  Activated partial thromboplastin time prolonged | 1 | 0 | 0 | 0 | 0
  Platelet count decreased | 0 | 0 | 1 | 0 | 0
  Blood fibrinogen decreased | 0 | 0 | 0 | 0 | 1
  Hepatic function abnormal | 0 | 1 | 1 | 0 | 0
  Alanine aminotransferase increased | 2 | 1 | 2 | 2 | 2
  Aspartate aminotransferase increased | 2 | 2 | 3 | 3 | 2
  Blood alkaline phosphatase increased | 0 | 2 | 1 | 2 | 2
  Blood bilirubin increased | 0 | 2 | 0 | 1 | 1
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 2 | 1
  Hyperthyroidism | 1 | 0 | 1 | 0 | 0
  Hypothyroidism | 0 | 0 | 0 | 4 | 0
  Blood thyroid stimulating hormone increased | 3 | 0 | 0 | 0 | 0
  Thyroxine free decreased | 1 | 0 | 0 | 0 | 0
  Tri-iodothyronine free decreased | 2 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormal Vital Signs and Physical Examinations Reported as TEAEs in Phase 2
Description: as for outcome 4
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Participants
  Atrial fibrillation | 1 | 1 | 1 | 0 | 0
  Bradycardia | 0 | 0 | 1 | 1 | 0
  Hypertension | 1 | 0 | 0 | 1 | 1
  Hypotension | 6 | 3 | 1 | 2 | 1
  Hypoxia | 2 | 0 | 1 | 0 | 0
  Pyrexia | 5 | 7 | 2 | 4 | 2
  Respiratory distress | 1 | 0 | 0 | 0 | 0
  Sinus tachycardia | 3 | 1 | 0 | 0 | 0
  Tachycardia | 1 | 0 | 1 | 1 | 0
  Weight decreased | 3 | 4 | 1 | 5 | 2

18. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms Reported as TEAEs in Phase 2
Description: as for outcome 5
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Participants
  Sinus tachycardia | 3 | 1 | 0 | 0 | 0
  Angina pectoris | 1 | 0 | 0 | 1 | 0
  Ventricular tachycardia | 1 | 0 | 1 | 0 | 0
  Tachycardia | 1 | 0 | 1 | 1 | 0
  Atrial fibrillation | 1 | 1 | 1 | 0 | 0
  Cardiac failure congestive | 1 | 0 | 0 | 0 | 0
  Atrial tachycardia | 0 | 1 | 0 | 0 | 0
  Bradycardia | 0 | 0 | 1 | 1 | 0
  Pericardial effusion | 0 | 0 | 1 | 0 | 0
  Cardiac failure | 0 | 0 | 0 | 0 | 1

19. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline in Phase 2
Description: as for outcome 6
Time Frame: Baseline (Day 1)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Participants
  ECOG 0 | 9 | 9 | 4 | 11 | 11
  ECOG 1 | 18 | 14 | 8 | 14 | 8

20. Secondary Outcome: Percentage of Participants With Disease Control at 16 Weeks in Phase 2
Description: The disease control rate at 16 weeks was defined as the percentage of participants who achieved a BOR of confirmed CR, confirmed PR, or had SD with duration of SD for a minimum duration of 110 days, following the date of randomization for Arm A, B, and C participants and the date of first dose of study drug for Arm D and E participants. The DC was defined as a BOR of confirmed CR, confirmed PR or SD per RECIST v1.1. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD on study.
Time Frame: From Day 1 up to 16 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Percentage of participants | 18.5 [6.3 to 38.1] | 12.5 [2.7 to 32.4] | 16.7 [2.1 to 48.4] | 28.0 [12.1 to 49.4] | 21.1 [6.1 to 45.6]

21. Secondary Outcome: Percentage of Participants With Disease Control at 24 Weeks in Phase 2
Description: The disease control rate at 24 weeks was defined as the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or had SD with duration of SD for a minimum duration of 166 days, following the date of randomization for Arm A, B, and C participants and the date of first dose of study drug for Arm D and E participants. The DC was defined as a BOR of confirmed CR, confirmed PR or SD per RECIST v1.1. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD on study.
Time Frame: From Day 1 up to 24 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Percentage of participants | 11.1 [2.4 to 29.2] | 0 [0.0 to 14.2] | 16.7 [2.1 to 48.4] | 12.0 [2.5 to 31.2] | 15.8 [3.4 to 39.6]

22. Secondary Outcome: Duration of Response (DoR) in Phase 2
Description: The DoR was defined as the time from the date of first documented response (CR or PR) until the first date of documented progression according to RECIST v1.1 that occurred subsequently after response or death due to any cause, whichever occurred first. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline. Kaplan Meier method was used to evaluate DoR.
Time Frame: From Day 1 up to End of the Treatment (EOT), 90 days post-EOT, every 3 months (Q3M) after Day 90 post-EOT up to 12 month post-EOT, and every 6 months after month 12 post-EOT (approximately up to 4 years and one month)
Population: As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received. Participants with OR were analyzed for the specified outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 3 | 0 | 1 | 1 | 3
Months | NA [2.0 to 22.4] — Median was not estimable because insufficient number of participants had events. |  | 4.6 [4.6 to 4.6] | 7.4 [7.4 to 7.4] | 3.1 [1.9 to 7.4]

23. Secondary Outcome: Time to Response (TTR) in Phase 2
Description: TTR: time from date of randomization of participants for Arm A, B, and C or date of first dose of study drug for Arm D and Arm E until first documented OR per RECIST v1.1. OR: BOR of confirmed CR or PR per RECIST v1.1. BOR: best response (CR, PR, SD, PD, and not evaluable) among all overall responses recorded from date of randomization/date of first dose of study drug until progression, or last evaluable disease assessment or discontinuation from the study, whichever occurred first. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in SOD of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD; PD: at least 20% increase in SOD of target lesions from smallest sum (at least 5mm), appearance of one or more new lesions, substantial worsening in non-target disease, increase in tumor burden leading to discontinuation of therapy. Kaplan Meier method used to evaluate TTR.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 3 | 0 | 1 | 1 | 3
Months | 1.9 [1.9 to 3.7] |  | 2.7 [2.7 to 2.7] | 7.2 [7.2 to 7.2] | 1.8 [1.7 to 1.8]

24. Secondary Outcome: Duration of Stable Disease in Phase 2
Description: The DSD was defined as the time from the date of randomization for Arm A, B, and C participants or the date of first dose of study drug for Arm D and Arm E participants until the first date of documented PD (per RECIST v1.1), or death due to any cause, whichever occurred first. PD is at least a 20% increase in sum of diameters of target lesions from smallest sum on study (at least 5 mm), appearance of one or more new lesions, substantial worsening in non-target disease, increase in tumor burden leading to discontinuation of therapy. Kaplan Meier method was used to evaluate DSD.
Time Frame: as for outcome 22
Population: as for outcome 10
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 4 | 3 | 1 | 6 | 1
Months | 3.5 [2.8 to 3.7] | 3.6 [3.5 to 4.3] | 7.7 [7.7 to 7.7] | 4.2 [3.5 to 7.2] | 3.5 [3.5 to 3.5]

25. Secondary Outcome: Median Best Percentage Change From Baseline of the Sum of Longest Diameters (SLD) of Target Lesions in Phase 2
Description: as for outcome 11
Time Frame: as for outcome 22
Population: As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received. Participants with any reduction in tumor size were analyzed for the specified outcome measure.
Measure: Median (Full Range); unit: mm
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 25 | 17 | 9 | 21 | 17
mm | 8.00 [-86.7 to 123.0] | 21.20 [-60.0 to 101.2] | -4.00 [-61.1 to 67.2] | 0.00 [-58.4 to 116.2] | 3.00 [-100.0 to 54.8]

26. Secondary Outcome: Progression Free Survival in Phase 2
Description: The PFS was defined as the time from the date of randomization for Arm A, B, and C participants or the date of first dose of study treatment for Arm D and E participants to the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1) or death due to any cause. PFS was censored at the date of their last evaluable tumor assessment. Kaplan Meier method was used to evaluate PFS.
Time Frame: as for outcome 22
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Months | 1.8 [1.6 to 2.8] | 1.6 [1.0 to 1.8] | 1.7 [0.8 to 7.3] | 1.8 [1.6 to 3.5] | 1.8 [1.6 to 1.9]

27. Secondary Outcome: Progression Free Survival at 9 Month (PFS-9) in Phase 2
Description: The PFS-9 is the 9-month progression-free survival rate, which was the percentage of participants who were progression free and alive at 9 months. PFS was defined as the time from the date of first dose of study drug for Arm A, B, C participants or the date of first dose of study drug for Arm D and E participants to the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1) or death due to any cause. PFS was censored at the date of their last evaluable tumor assessment. Kaplan Meier method was used to evaluate PFS.
Time Frame: From Day 1 up to 9 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Percentage of participants | 12.1 [3.1 to 27.9] | NA [NA to NA] — No participants were progression free at 9 months. | NA [NA to NA] — No participants were progression free at 9 months. | 4.2 [0.3 to 17.6] | 5.3 [0.4 to 21.4]

28. Secondary Outcome: Overall Survival (OS) in Phase 2
Description: The OS was defined as the time from date of randomization for Arm A, B, and C participants or the date of first dose of study drug for Arm D and Arm E participants until death due to any cause. OS was censored at last known alive date. Kaplan Meier method was used to evaluate OS. Kaplan Meier method was used to evaluate OS.
Time Frame: as for outcome 22
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Months | 9.2 [1.6 to 32.0] | 3.4 [0.8 to 9.5] | 7.7 [0.8 to 33.8] | 10.7 [1.0 to 30.7] | 7.0 [0.6 to 18.8]

29. Secondary Outcome: Overall Survival at 12 Months in Phase 2
Description: The OS was defined as the time from date of randomization for Arm A, B, and C participants or the date of first dose of study drug for Arm D and Arm E participants until 12 months. OS was censored at last known alive date. Kaplan Meier method was used to evaluate OS. Kaplan Meier method was used to evaluate OS and 95% confidence interval.
Time Frame: From Day 1 up to 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Percentage of participants | 37.0 [19.6 to 54.6] | NA [NA to NA] — No participants were alive at 12 months. | 13.1 [0.7 to 43.6] | 40.7 [20.2 to 60.3] | 29.2 [10.9 to 50.5]

30. Secondary Outcome: Percentage of Participants With Objective Response With Positive Interferon Gamma (IFN-γ) Gene Expression in Phase 2
Description: Percentage of participants with OR with positive IFN-γ gene expression is reported. OR: BOR of confirmed CR or PR per RECIST v1.1. BOR: best response (CR, PR, SD, PD, and not evaluable) among all overall responses recorded from date of randomization for Arm A, B, C participants or date of first dose of study drug for Arms D, E participants until progression, or last evaluable disease assessment or discontinuation from the study, whichever occurred first. CR: disappearance of all target/non-target lesions; PR: at least 30% decrease in sum of diameters (SOD) of target lesions from baseline; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD from smallest SOD on study; PD: at least 20% increase in SOD of target lesions from smallest sum on study (at least 5mm), appearance of one or more new lesions, substantial worsening in non-target disease, increase in tumor burden leading to discontinuation of therapy.
Time Frame: Day 1 through Day 30 post EOT (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percenatge of Participants
Arm/Group | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 19
Percenatge of Participants | 15.8 [3.4 to 39.6]

31. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 6 Month With Positive IFN-γ Gene Expression in Phase 2
Description: Percentage of participants with PFS at 6 month with positive IFN-γ gene expression is reported. The PFS-6 is the 6-month progression-free survival rate, which was the percentage of participants who were progression free and alive at 6 months. PFS was defined as the time from the date of first dose of study drug for Arm A, B, and C participants or the date of first dose of study drug for Arm D and Arm E participants to the earlier of the dates of the first objective documentation of radiographic disease progression (per RECIST v1.1) or death due to any cause. PFS was censored at the date of their last evaluable tumor assessment. Kaplan Meier method was used to evaluate PFS-6.
Time Frame: Day 1 through Day 30 post EOT (approximately 4 years and one month)
Population: As-treated population included all participants who received any study drug and analyzed according to the treatment they actually received. Only those participants were analyzed who were at risk at 6 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 1
Percentage of Participants | 5.3 [0.4 to 21.4]

32. Secondary Outcome: Percentage of Participants With Objective Response in Phase 2 by Programmed Death-ligand (PD-L1) Status
Description: Percentage of participants with objective response in Phase 2 by programmed death-ligand (PD-L1) status is reported. PD-L1 is a protein that may be found on some normal cells and in higher-than-normal amounts on some types of cancer cells. It plays a role in regulating the immune response against some types of cancers and therefore, is the target for some anticancer drugs. PD-L1 status was based on the percentage of tumor cells from baseline tumor tissue samples with PD-L1 membrane staining: PD-L1 high if >= 1% tumor cells (better response), PD-L1 low/neg if < 1% tumor cells (low response).
Time Frame: Day 1 through Day 30 post EOT (approximately 4 years and one month)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
Number analyzed (Participants) | 27 | 24 | 12 | 25 | 19
Percentage of participants
  PD-L1 high: number analyzed (Participants) | 15 | 11 | 7 | 5 | 9
  PD-L1 high | 13.3 [1.7 to 40.5] | 0 [0.0 to 28.5] | 0 [0.0 to 41.0] | 0 [0.0 to 52.2] | 33.3 [7.5 to 70.1]
  PD-L1 low/negative: number analyzed (Participants) | 9 | 9 | 4 | 15 | 4
  PD-L1 low/negative | 11.1 [0.3 to 48.2] | 0 [0.0 to 33.6] | 25.0 [0.6 to 80.6] | 0 [0.0 to 21.8] | 0 [0.0 to 60.2]

ADVERSE EVENTS:
Time Frame: Day 1 up to 90 days after the last dose (approximately 4 years and one month)
Arm/Group | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W) | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm B-M10 mg/kg (Q2W) | Phase 2 Arm C-T10 mg/kg (Q4W) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W)
All-Cause Mortality (participants affected / at risk) | 6/6 | 23/27 | 21/24 | 7/12 | 21/25 | 13/19
Serious Adverse Events (participants affected / at risk) | 2/6 | 14/27 | 16/24 | 10/12 | 15/25 | 12/19
Other Adverse Events (participants affected / at risk) | 6/6 | 27/27 | 22/24 | 12/12 | 22/25 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W) (N=6) | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (N=27) | Phase 2 Arm B-M10 mg/kg (Q2W) (N=24) | Phase 2 Arm C-T10 mg/kg (Q4W) (N=12) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (N=25) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b-M20 mg/kg (Q4W) + T 1 mg/kg (Q4W) Fw M10 mg/kg (Q2W) (N=6) | Phase 2 Arm A-(M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (N=27) | Phase 2 Arm B-M10 mg/kg (Q2W) (N=24) | Phase 2 Arm C-T10 mg/kg (Q4W) (N=12) | Phase 2 Arm D-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (N=25) | Phase 2 Arm E-M20 mg/kg (Q4W) + T1 mg/kg Fw M10 mg/kg (Q2W) (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 9 (16) | 3 (6) | 3 (8) | 8 (13) | 4 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (7) | 3 (3) | 4 (4) | 5 (5) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 4 (5) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 9 (10) | 5 (6) | 4 (4) | 3 (6) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 9 (12) | 3 (4) | 5 (6) | 4 (8) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 2 (8) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (20) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (11) | 5 (6) | 4 (11) | 8 (12) | 6 (8)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (7) | 3 (3) | 3 (8) | 8 (15) | 4 (10)
Asthenia (General disorders) | 0 (0) | 2 (5) | 6 (6) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 11 (31) | 6 (6) | 5 (14) | 9 (12) | 5 (6)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 6 (7) | 1 (1) | 3 (5) | 5 (6) | 4 (4)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 5 (7) | 6 (7) | 2 (5) | 3 (6) | 2 (3)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (5) | 2 (3) | 2 (2) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (4) | 2 (8) | 3 (5) | 3 (3) | 2 (2)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 3 (9) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (3) | 1 (1) | 2 (3) | 1 (1) | 3 (8)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (13) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 5 (5) | 2 (3)
Weight increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 10 (28) | 8 (9) | 5 (14) | 9 (15) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (14) | 1 (3) | 0 (0) | 1 (2) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (11) | 1 (1) | 3 (3) | 5 (10) | 3 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 3 (3) | 1 (3) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 2 (4) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 3 (3) | 1 (2) | 2 (2) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 5 (8) | 1 (1) | 0 (0) | 2 (5) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (14) | 2 (2) | 3 (3) | 6 (11) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 3 (7) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 7 (10) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital erosion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 2 (2) | 1 (2) | 2 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 10 (15) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (9) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (21) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (8) | 0 (0) | 5 (8) | 6 (6) | 3 (5)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 5 (6) | 2 (2) | 1 (1) | 3 (4) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT02340975/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT02340975/SAP_001.pdf